CLINICAL TRIAL: NCT06763757
Title: Art Application and Transformation on Solitary Seniors.
Brief Title: Art Therapy for Enhancing Well-Being in Solitary Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Yunlin University of Science and Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202410001RINA
Record Dates: First submitted 2024-12-27; First posted 2025-01-08 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Mental Health; Quality of Life; Emotional Well-being; Loneliness
Keywords: Occupational Therapy; Solitary Older Adults; Mental Health; Quality of Life; Art Therapy
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy Intervention Group (Experimental): Participants in the experimental group will attend 12 weekly art therapy sessions, each lasting 90 minutes. These sessions are designed to enhance emotional well-being, foster self-expression, and improve interpersonal connections through guided art activities. The program includes creating art, observing and discussing art pieces, and engaging in reflective exercises to explore personal emotions and experiences. Each session is structured to build upon the previous ones, beginning with activities to establish trust and comfort, progressing to deeper emotional exploration, and culminating in a final creative project. The sessions are led by trained facilitators and supervised by licensed occupational therapists. Evaluations will be conducted before and after the 12-week program using the Taiwanese version of the WHO Quality of Life-BREF (WHOQOL-BREF) and the Beck Depression Inventory (BDI) to assess changes in mental health and quality of life
  Interventions: Behavioral: Art Therapy Program
- No Intervention Control Group (No Intervention): Participants in the control group will not receive any intervention during the study period and will continue with their usual daily routines. They will complete two evaluations: one at baseline before the start of the study and another after 12 weeks. These evaluations will use the Taiwanese version of the WHO Quality of Life-BREF (WHOQOL-BREF) and the Beck Depression Inventory (BDI) to measure mental health and quality of life. The data collected will serve as a comparison to determine the effectiveness of the art therapy intervention in the experimental group.

INTERVENTIONS:
Behavioral: Art Therapy Program — The Art Therapy Program consists of 12 weekly group sessions, each lasting 90 minutes, designed to improve emotional well-being and quality of life in solitary older adults. Participants engage in structured activities that include creating art (e.g., drawing and painting), observing and interpreting art pieces, and reflective discussions to explore personal emotions and experiences. The sessions are led by trained facilitators under the supervision of licensed occupational therapists. This intervention follows a thematic progression: initial sessions focus on building trust and self-expression, mid-sessions deepen emotional awareness, and final sessions culminate in a creative project reflecting the participant's personal growth. Unlike other interventions, this program is tailored specifically for older adults living alone, addressing their unique challenges of isolation and reduced social interaction.
  Arms: Art Therapy Intervention Group

SUMMARY:
This study explores the impact of art therapy on mental health and quality of life among solitary older adults. Participants will be randomly assigned to one of two groups: an experimental group receiving art therapy sessions or a control group with no intervention. The art therapy program includes 12 weekly sessions lasting 90 minutes each, focusing on creative expression, observation of art, and reflective discussions. These activities are designed to enhance emotional well-being, reduce depressive symptoms, and foster interpersonal connections.

Both groups will undergo evaluations before and after the 12-week study period. The assessments will include the Taiwanese version of the WHO Quality of Life-BREF (WHOQOL-BREF) and the Beck Depression Inventory (BDI) to measure changes in psychological health and life satisfaction. The findings aim to demonstrate the feasibility and benefits of art therapy as a non-pharmacological intervention for improving the well-being of solitary older adults.

DETAILED DESCRIPTION:
This study explores the effects of art therapy on mental health and quality of life among solitary older adults. The research examines whether engaging in creative activities can reduce loneliness, enhance emotional well-being, and improve life satisfaction in this vulnerable population.

Living alone presents significant emotional and social challenges for older adults, increasing the risk of depression, isolation, and reduced quality of life. Art therapy, which combines creativity with emotional expression, offers a promising, non-invasive approach to address these issues. While its benefits are documented in other populations, its specific impact on solitary older adults is not fully understood. This study aims to provide evidence on how structured art therapy programs can support this group.

This study investigates the effects of art therapy on the mental health and quality of life of solitary older adults. Solitary living often increases the risk of depression, isolation, and reduced life satisfaction, making non-pharmacological interventions like art therapy a promising approach to address these challenges. This randomized controlled trial evaluates the feasibility and effectiveness of a structured art therapy program in enhancing psychological well-being and overall quality of life.

Participants will be randomly assigned to either the experimental group or the control group. The experimental group will attend 12 weekly art therapy sessions, each lasting 90 minutes. These sessions include hands-on art creation, discussions on art observation and interpretation, and reflective exercises to explore personal emotions and experiences. The program is designed to foster self-expression, enhance interpersonal connections, and promote emotional resilience. The control group will not receive any intervention and will continue their usual daily routines. Both groups will complete standardized assessments before and after the 12-week study period.

Evaluations will use the Taiwanese version of the WHO Quality of Life-BREF (WHOQOL-BREF) and the Beck Depression Inventory (BDI) to measure changes in psychological health and life satisfaction. The data collected will compare outcomes between the two groups to determine the impact of the art therapy intervention.

This study has been reviewed and approved by the Institutional Review Board (IRB) of the National Taiwan University Hospital Yunlin Branch. Written informed consent will be obtained from all participants, and their data will be securely stored and de-identified to ensure confidentiality. The findings aim to provide valuable insights into the use of art therapy as a scalable, non-pharmacological intervention for improving the mental health and quality of life of solitary older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older.
2. Living alone.
3. Mini-Mental State Examination (MMSE) score between 24 and 30, indicating no significant cognitive impairment.
4. Capable of providing informed consent.
5. Physically able to participate in art-related activities such as drawing or painting.
6. Not currently undergoing psychiatric medication treatment for conditions such as depression, anxiety, schizophrenia, or bipolar disorder.

Exclusion Criteria:

1. Recent major life events (e.g., bereavement, severe illness) that could interfere with study participation.
2. History of brain injury or severe psychiatric conditions, such as schizophrenia or major depressive disorder requiring hospitalization.
3. Physical disabilities or motor impairments that prevent participation in art activities.
4. Participation in similar art therapy studies within the past 6 months.
5. Strong aversion or resistance to art therapy activities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life (WHOQOL-BREF) | Baseline (pre-intervention) and 12 weeks (post-intervention).
  The primary outcome is the change in quality of life scores, as measured by the Taiwanese version of the WHO Quality of Life Questionnaire-BREF (WHOQOL-BREF). This tool evaluates quality of life across four domains: physical health, psychological well-being, social relationships, and environmental factors. Each domain is scored independently, with scores ranging from 0 to 100. Higher scores indicate better quality of life, reflecting positive perceptions in that domain.

SECONDARY OUTCOMES:
Change in Depressive Symptoms (BDI) | Baseline (pre-intervention) and 12 weeks (post-intervention).
  The Beck Depression Inventory (BDI) is a self-reported questionnaire used to measure the severity of depressive symptoms. It consists of 21 items, each scored on a scale of 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate more severe depressive symptoms. The BDI is widely validated and commonly used in both clinical and research settings to assess changes in depression severity over time, making it ideal for evaluating the impact of interventions on mental health outcomes.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the study will be shared to support secondary research. This includes demographic data, baseline characteristics, and outcome measures (e.g., scores from the WHOQOL-BREF and Beck Depression Inventory). The shared data will exclude direct identifiers to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP
Time Frame: The de-identified individual participant data (IPD) and supporting information will be available starting 6 months after the publication of the primary study findings. The data will remain accessible for a period of 5 years following the initial release.
Access Criteria: De-identified individual participant data (IPD) and supporting information, including the study protocol, statistical analysis plan, and informed consent form, will be accessible to qualified researchers who submit a formal data access request. The request must include a detailed research proposal outlining the intended use of the data, methods of analysis, and publication plans. Proposals will be reviewed and approved by the principal investigator and the Institutional Review Board (IRB) to ensure ethical and scientific validity. Approved researchers will be required to sign a data-sharing agreement to ensure compliance with data use policies. The data and documents will be shared through a secure external repository, with access granted on a case-by-case basis.

REFERENCES:
- [Derived] Tsai PC, Chou WH, Liao SY. A randomized controlled trial study of a life review art intervention for older adults living alone. Front Psychol. 2025 Nov 19;16:1669119. doi: 10.3389/fpsyg.2025.1669119. eCollection 2025. PMID 41346530